CLINICAL TRIAL: NCT05373589
Title: Effect of Pressure Support Ventilation During Anesthetic Emergence on Postoperative Atelectasis in Infant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 4-2022-0119
Record Dates: First submitted 2022-04-29; First posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Infants Aged 0 Days to 13 Months Scheduled for Elective Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group C (Experimental)
  Interventions: Other: conventional ventilation, group C
- group PS (Experimental)
  Interventions: Other: pressure support, group PS

INTERVENTIONS:
Other: conventional ventilation, group C — In the conventional ventilation group, after stopping the administration of the inhalation gas, the emergence process is performed by the anesthesiologist assigned to the room. Basically, until spontaneous respiration of the patient is restored, an anesthesiologist can assist respiration by intermittent manual assistance if necessary.
  Arms: group C
Other: pressure support, group PS — In the pressure support group, after stopping the administration of the inhalation gas, switch to the pressure support mode at the emergence period. PEEP 5cmH20 is applied, and the safety backup ventilation rate is set to 12 breaths/min. The flow trigger is set to 1L/min, and the degree of support is made to be 7-8ml of the predicted body weight, and is decreased as the patient's spontaneous breathing is restored.
  Arms: group PS

SUMMARY:
Atelectasis occurs in patients of all ages who receive mechanical ventilation under general anesthesia, and although fatal cases are rare, it is known as a cause of postoperative hypoxia or fever. In pediatric patients, it has a particularly high incidence of 68-100%, and the incidence is inversely proportional to age. Pediatric patients,compared to adults, have a small capacity for functional residual capacity while a high metabolic demand, making them fundamentally vulnerable to hypoxia. Increased atelectasis during anesthesia causes hypoxia not only during anesthesia but also during recovery after anesthesia. Therefore, it is important to establish and apply a strategy to minimize the occurrence of atelectasis during mechanical ventilation under general anesthesia in pediatric patients. The aim of this study is to investigate whether pressure support ventilation at emergence period could reduce the incidence of postoperative atelectasis in infants undergoing surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. infant patients aged 0 day to 13 month
2. American Society of Anesthesiologists (ASA) classification 1~2 who are scheduled for elective surgery under general anesthesia

Exclusion Criteria:

1. patients with symptomatic bronchopulmonary dysplasia
2. patients with uncorrected congenital heart or pulmonary disease
3. Hemodynamically unstable requiring preoperative vasopressor administration
4. fever (>37.5°) or URI symptoms on the day of surgery

Ages: 0 Years to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 136 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Frequency of atelectasis | Within 5 minutes of arriving at the recovery room
  Immediately after arriving at the recovery room, lung ultrasound is performed to check for atelectasis.

SECONDARY OUTCOMES:
Frequency of atelectasis | After 30 minutes of stay in the recovery room
  After 30 minutes of staying in the recovery room, lung ultrasound was performed to check for atelectasis.
scoring of atelectasis | at the time of admission and after 30 minutes of stay in the recovery room
  Perform atelectasis scoring on 12 parts of the lung
Frequency of desatuation | at the time of admission and after 30 minutes of stay in the recovery room
  Check the frequency of desaturation (<95%) during the stay in the recovery room.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No